CLINICAL TRIAL: NCT00901069
Title: Azacitidine With Rituximab, Vincristine, and Cyclophosphamide in Refractory Lymphoma: A Phase I Trial
Brief Title: Azacitidine With Rituximab, Vincristine, and Cyclophosphamide in Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shams Shakil (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Shams Shakil, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-NHL-06-UK/CC; NCT00589160 (obsolete NCT alias)
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Azacitidine; Rituximab; Vincristine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine (Other)
  Interventions: Drug: Azacitidine with rituximab, vincristine, and cyclophosphamide

INTERVENTIONS:
Drug: Azacitidine with rituximab, vincristine, and cyclophosphamide — Azacitidine cycle days 1-5 Cyclophosphamide cycle days 6-9 Vincristine cycle day 8 Rituximab cycle day 8 Rituximab is only for those patients with CD20+ lymphoma. Azacitidine 25 mg/m2^ Azacitidine 50 mg/m2^ Azacitidine 75 mg/m2^ Azacitidine 100 mg/m2^

SUMMARY:
This is a phase I, prospective, open label, dose escalation study of azacitidine in combination with rituximab, vincristine, and cyclophosphamide for the treatment of refractory lymphoma. The investigators expect to enroll 12-24 patients in this trial over a 2 year accrual period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or their authorized legally acceptable representative must consent to be in the study and must have signed and dated an approved consent form which conforms to federal and institutional guidelines.
2. Age ≥ 18 years and without a maximum age.
3. All patients of reproductive potential should not plan on conceiving children during the treatment program and must agree to use a medically accepted form of contraception.
4. Women of childbearing potential must have a negative serum pregnancy test within 2 weeks of beginning treatment.
5. Patients must have relapsed lymphoma.
6. ECOG performance status of 2 or better.

Exclusion Criteria:

1. Pregnant or breast-feeding at the time of proposed study entry
2. Clinical AIDS or ARS or known positive HIV serology
3. History of malignant neoplasm, other than lymphoma, treated within two years prior to study entry (other than non-melanoma skin cancer or in situ cervical cancer) or where there is current evidence of recurrent or metastatic disease
4. Psychiatric or additive disorders that would preclude obtaining informed consent
5. Serum bilirubin > 1.5 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these are attributed to active hemolysis
6. Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels > 2 times ULN
7. Serum creatinine levels > 1.5 times ULN
8. Platelets < 75,000/mm3
9. Absolute neutrophil count < 1500/mm3
10. Active infection including viral hepatitis
11. Known or suspected hypersensitivity to mannitol, azacitidine, or rituximab
12. Grade 3 or 4 neuropathy
13. Advanced hepatic tumors
14. Uncompensated heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determine the maximal tolerated dose (MTD) of azacitidine in combination with rituximab, vincristine, and cyclophosphamide in patients with lymphoma | Eight 21 day cycles

CONTACTS AND LOCATIONS:
Overall Officials: Shams Shakil, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States